CLINICAL TRIAL: NCT03992950
Title: Effectiveness of Cricoid and Paratracheal Pressures for Occluding Esophagus in Anesthetized and Paralyzed Patients During the Induction of Anesthesia
Brief Title: Effectiveness of Cricoid and Paratracheal Pressures for Occluding Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P2019-195
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricoid pressure (Experimental): Cricoid pressure is applied in the anesthetized state and during video laryngoscopy
  Interventions: Other: Maneuvers for occluding esophagus
- Paratracheal pressure (Experimental): Paratracheal pressure is applied in the anesthetized state and during video laryngoscopy
  Interventions: Other: Maneuvers for occluding esophagus

INTERVENTIONS:
Other: Maneuvers for occluding esophagus — Cricoid pressure: pressure on the cricoid ring Paratracheal pressure: pressure on the left paratracheal region below the cricoid level

SUMMARY:
Comparing the effects of 'Cricoid pressure' or 'Paratracheal pressure' during direct laryngoscopy

DETAILED DESCRIPTION:
The effectiveness of cricoid pressure and paratracheal pressure for occluding esophagus during direct and video laryngoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Who would be scheduled any surgery under general anesthesia and agree with the purpose of the study

Exclusion Criteria:

* Risk of aspiration
* History of esophageal surgery
* Diseases or anatomical abnormalities of the neck, larynx, pharynx or esophagus
* Known or predicted difficult airway.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Occlusion of the esophagus | During 1 minute under videolaryngoscopy
  Occlusion of the esophagus is checked with the application of cricoid and paratracheal pressures using esophageal stethoscope. If the esophageal stethoscope is not advanced into the esophagus, it is considered 'occlusion'.

SECONDARY OUTCOMES:
Outer diameter of the esophagus | During 1 minute after injection of anesthetics during induction of anesthesia
  Outer diameter of the esophagus is measured using ultrasound before and after the application of cricoid and paratracheal pressures.
Position of the oesophageal entrance relative to the glottis | During 1 minute after injection of anesthetics during induction of anesthesia and during videolaryngoscopy
  Position of the oesophageal entrance relative to the glottis is evaluated.
Position of the upper oesophagus relative to the trachea | During 1 minute after injection of anesthetics during induction of anesthesia and during videolaryngoscopy
  Position of the upper oesophagus relative to the trachea trachea is evaluated.
The best laryngeal view | Before and after the application of cricoid and paratracheal force during videolaryngoscopy
  The best laryngeal view is evaluated using the percentage of glottis opening (POGO) score, ranging from 0% to 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Chang JE, Won D, Lee JM, Kim TK, Kim MJ, Min SW, Hwang JY. Effectiveness of Cricoid and Paratracheal Pressures in Occluding the Upper Esophagus Through Induction of Anesthesia and Videolaryngoscopy: A Randomized, Crossover Study. Anesth Analg. 2022 Nov 1;135(5):1064-1072. doi: 10.1213/ANE.0000000000006154. Epub 2022 Aug 1. PMID 35913721